CLINICAL TRIAL: NCT06732726
Title: Assessment of the Padua Prediction Score for Venous Thromboembolism Risk Stratification in Thoracic Surgery Patients: Insights From a Single-Center Cohort Study in Iraq
Brief Title: Padua Prediction Score for VTE Risk in Thoracic Surgery Patients
Acronym: DVT
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241210; 008 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: DVT - Deep Vein Thrombosis; VTE (Venous Thromboembolism)
Keywords: Padua Prediction Score (PPS)
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this observational study is to assess the predictive accuracy of the Padua Prediction Score (PPS) for venous thromboembolism (VTE) risk in thoracic surgery patients.

The study aims to answer the following question:

Does the PPS provide a more accurate prediction of VTE risk?

Participants will:

Have their VTE risk assessed using the PPS during their hospital admission.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a significant cause of morbidity and mortality, comprising conditions like deep vein thrombosis (DVT) and pulmonary embolism (PE). Hospitalized patients are particularly vulnerable to VTE due to factors such as prolonged immobility, surgical procedures, and preexisting comorbidities.

To address this risk, tools like the Padua Prediction Score (PPS) have been developed. PPS is a validated scoring system that uses clinical and demographic criteria to categorize patients as high- or low-risk for VTE, allowing healthcare providers to tailor prophylactic measures accordingly. Although the Padua Prediction Score has been increasingly adopted in various healthcare settings, its applicability in Iraq remains understudied. There is limited local data on the prevalence of VTE, risk assessment practices and adherence to prophylaxis protocols, leaving a clear gap in the literature. This study aims to explore the utility and predictive accuracy of the Padua Prediction Score in the Iraqi healthcare context. By addressing this gap, the findings could help refine VTE prevention strategies, improve resource allocation, and ultimately reduce complications associated with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone preoperative Padua Prediction Score assessment.
* Inpatients with a hospital stay over 3 days
* Written informed consent obtained from patients or their legal guardians.
* Availability for postoperative follow-up to assess outcomes like LEVT development or related complications.

Exclusion Criteria:

* Preexisting LEVT or pulmonary embolism.
* Severe Coagulopathy: Patients with inherited or acquired bleeding disorders (e.g., hemophilia, advanced liver disease).
* receiving any anticoagulation therapy for any reason.
* patients who did not undergo a postoperative D-dimer test.
* Incomplete Data: missing essential clinical or laboratory data.
* Pregnancy: pregnant women or those within six weeks postpartum.
* Noncompliance: Patients unwilling or unable to adhere to study follow-up protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will focus on adult patients undergoing thoracic surgery at a single center in Iraq.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Venous Thromboembolism (VTE) Episodes in Patients | In-Hospital Phase (average of 10 days through discharge); Post-Discharge Follow-Up: Day 7, Day 15, and Day 30
  symptomatic or asymptomatic, confirmed by instrumental diagnostics.
Padua Prediction Score | Day 1 preoperative (one day prior to surgery)
  A total score that ranges from 0 to 20. 4 or higher indicates a significant likelihood of developing VTE.

SECONDARY OUTCOMES:
Incidence of Symptomatic Pulmonary Embolism in Patients | In-Hospital Phase (average of 10 days through discharge); Post-Discharge Follow-Up: Day 7, Day 15, and Day 30
  symptomatic pulmonary embolism confirmed by perfusion isotope scanning or CT pulmonary angiography.
Rate of Recurrent Deep Vein Thrombosis (DVT) in Patients | Post-Discharge Follow-Up: Day 7, Day 15, and Day 30
  A new episode of deep vein thrombosis occurs after the initial diagnosis with clinical symptoms (such as leg pain, swelling, redness, or tenderness) and is confirmed through instrumental diagnostics (e.g., ultrasound, CT venography, MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Yaser aamer Eisa Alhaibi, Assistant professor, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Kadhimiya, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Yami MS, Silva MA, Donovan JL, Kanaan AO. Venous thromboembolism prophylaxis in medically ill patients: a mixed treatment comparison meta-analysis. J Thromb Thrombolysis. 2018 Jan;45(1):36-47. doi: 10.1007/s11239-017-1562-5. PMID 29043538
- [Result] Barbar S, Noventa F, Rossetto V, Ferrari A, Brandolin B, Perlati M, De Bon E, Tormene D, Pagnan A, Prandoni P. A risk assessment model for the identification of hospitalized medical patients at risk for venous thromboembolism: the Padua Prediction Score. J Thromb Haemost. 2010 Nov;8(11):2450-7. doi: 10.1111/j.1538-7836.2010.04044.x. PMID 20738765